CLINICAL TRIAL: NCT02722044
Title: An Open-label Single-arm Multicenter Study to Evaluate Usability of a Subcutaneous (SC) Autoinjector (AI) for a Proposed Adalimumab Biosimilar (M923) in Subjects With Moderate to Severe Rheumatoid Arthritis (RA)
Brief Title: Usability of an AI for M923 in Subjects With Moderate to Severe RA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 911502
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Study Participants (Experimental): All study participants to receive M923 administered via a subcutaneous auto-injector (AI)
  Interventions: Biological: M923; Device: Autoinjector

INTERVENTIONS:
Biological: M923 — Recombinant human immunoglobulin G subclass 1 (IgG1) monoclonal antibody specific for human tumor necrosis factor-alpha (TNF-α)
  Other Names: Adalimumab
Device: Autoinjector — Subcutaneous administration

SUMMARY:
The purpose of this study is to evaluate the usability of an auto-injector (AI) for the delivery of M923 in patients with rheumatoid arthritis (RA)

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years old at the time of Screening
2. Able to understand and communicate with the Investigator and comply with the requirements of the study, and must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed study consent according to local laws and regulations.
3. RA diagnosed for at least 6 months before Screening
4. Meets classification criteria for rheumatoid arthritis (RA) by 2010 American College of Rheumatology/European League Against Rheumatism criteria
5. Active disease at Screening and Baseline
6. Participants must have at least 1 documented swollen and/or tender joint in their hand or wrist of the dominant hand as assessed by the Investigator or designated assessor
7. Must be willing and able to attempt self-administration of subcutaneous (SC) injection(s)
8. Male participants and their female partners must be willing to comply with the contraception restrictions for this study from the time of the first administration of investigational product (IP) until 3 months after the last dose.
9. Female participants must have a negative pregnancy test at screening and on admission to the clinic, and must not be lactating and must be using an acceptable method of contraception throughout the study and for 3 months after the last dose, or be of non-childbearing potential. Non-pregnant female partners of male participants who are of childbearing potential should use an effective form of contraception.

Exclusion Criteria:

1. Prior use of systemic tumor necrosis factor (TNF) inhibitor therapy.
2. Prior use of rituximab
3. Prior use of abatacept, tocilizumab and tofacitinib within 4 weeks prior to Screening
4. Current use of a conventional disease modifying anti-rheumatic drugs (DMARD) other than the following: methotrexate orally (≤25 mg/day), hydroxychloroquine (≤400 mg/day) or sulfasalazine (≤3 g/day)) at a stable dose for at least 4 weeks prior to Screening. If discontinued, methotrexate, hydroxychloroquine, and sulfasalazine must have been discontinued at least 4 weeks prior to Baseline. No other conventional DMARDs are permitted and no combination therapy is permitted.
5. Prior use of cytotoxic or alkylating agents or immunosuppressants must have been discontinued for at least 90 days prior to Baseline
6. Current use of oral corticosteroids at a dose >10 mg/day prednisone or equivalent or change of dose within 2 weeks prior to Screening
7. Current use of more than 1 nonsteroidal anti-inflammatory drug.
8. Prior use of injectable corticosteroids (intramuscular [IM], intra-articular [IA], or intravenous [IV]) within 6 weeks prior to Baseline
9. Prior or current use of other self-injected drugs, eg, insulin
10. All other prior non-RA concomitant treatments must be on a stable dose for at least 4 weeks before Baseline
11. Meets Class IV Steinbrocker criteria for disability/activities of daily living
12. Laboratory abnormalities at Screening deemed clinically significant by the Investigator and/or Sponsor.
13. Presence of fibromyalgia, another autoimmune rheumatologic illness or inflammatory arthritis, eg, systemic lupus erythematosus, gout. The presence of secondary Sjogren's syndrome is permitted.
14. Joint surgery within the last 8 weeks prior to Screening
15. Severe, progressive, or uncontrolled renal, hepatic, metabolic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac or neurologic disease, including pleural effusions or ascites, which in the opinion of the Investigator would preclude the participant from adhering to or completing the study or where participation in the study exposes the participant to unfavorable benefit/risk
16. History or presence of signs and/or symptoms or a diagnosis of a demyelinating disorder
17. History or presence of Class III or IV New York Heart Association congestive heart failure
18. History or presence of symptoms suggestive of lymphoproliferative disorders, lymphoma, leukemia, myeloproliferative disorders, or multiple myeloma
19. Existing malignancy or history of any malignancy except adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ, with no more than 3 lifetime basal cell or squamous cell carcinomas
20. Chronic infections, recurrent infections (3 or more of the same infection requiring anti-infective treatment in any rolling 12-month period); any recent infection (ie, in the last 30 days) requiring hospitalization or any infection requiring parenteral anti-infective therapy within 30 days or oral infective therapies within 14 days of Baseline; herpes zoster within 6 months of Baseline or more than 2 lifetime episodes of herpes zoster; or history of systemic fungal infection or opportunistic infection (eg, coccidioidomycosis, histoplasmosis, toxoplasmosis)
21. History or presence of human immunodeficiency virus (HIV), Hepatitis B or C virus
22. History of active tuberculosis (TB) or untreated or inadequately treated latent TB.
23. Participant has been exposed to an investigational product (IP) within 30 days (or 5 half-lives) prior to enrollment, whichever is longer, or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
24. Participant is a family member or employee of the Investigator or Baxalta or its partners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Caminis, MD, Study Director — Baxalta US Inc., now part of Shire
Locations (7):
- United States (7):
  - Henry Ford Health System, Detroit, Michigan
  - Medication Management, LLC, Greensboro, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, PC, Duncansville, Pennsylvania
  - Austin Regional Clinic, PA, Austin, Texas
  - Accurate Clinical Management, Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 participants were screened, and 33 participants were enrolled in the study.
Groups:
- M923 40 mg: Participants self-administered 40 milligrams (mg) of M923 every 2 weeks, as a subcutaneous injection using an auto-injector, for up to a maximum of 32 weeks.
Period: Overall Study
Arm/Group | M923 40 mg
Started | 33
Completed | 28
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Did Not Meet Criteria at Week 14 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received study medication
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Usability of the Auto-injector (AI) at Week 4
Description: The primary usability measure was the participant rating captured in the PRE- and POST-Self-injection Assessment Questionnaire (SIAQ) modules at Week 4. The PRE-SIAQ module is a 7-item questionnaire that investigates feelings about injections, self-confidence (regarding self-administration), and satisfaction with self-injection. The POST-SIAQ module is a 27-item questionnaire that assesses feelings about injections, self-image, self-confidence (regarding self-administration), pain and skin reactions during or after injection (injection-site reactions), ease of use of the self-injection device, and satisfaction with self-injection. Participants rated each item of the SIAQ on a 5-point (or 6-point) semantic Likert-type scale, where a score of 1 corresponds to a participant's worst experience and a score of 5 (or 6) corresponds to a participant's best experience. Item scores were transformed to obtain a score ranging from 0 (worst experience) to 10 (best experience) for each item.
Time Frame: Week 4
Population: Usability Analysis Set: all participants in the Safety Analysis Set who had usability measurements at Week 4 and who did not have any deviations from the protocol deemed significant enough for exclusion from the usability analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Scores on a scale
  Feelings about injections: PRE | 8.15 (2.049)
  Feelings about injections: POST | 8.17 (1.930)
  Self-image: POST | 9.27 (2.061)
  Self-confidence: PRE | 8.12 (2.183)
  Self-confidence: POST | 8.39 (2.287)
  Pain/skin reactions during/after injection: POST | 9.33 (0.630)
  Pain during/after injection: POST | 8.76 (1.234)
  Skin reactions: POST | 9.90 (0.301)
  Ease of use of the AI: POST | 8.72 (2.072)
  Satisfaction with self-injection: PRE | 8.39 (1.887)
  Satisfaction with self-injection: POST | 8.89 (1.369)

2. Secondary Outcome: Number of Participants With Successful Injections as Assessed by the Observer at Week 4
Description: Observers assessed usability by using a self-injection checklist. Self-injection assessment was coded as successful if categories P7 (removed protective needle cap from auto-injector), P10 (press down on auto-injector to insert the needle into the skin), and P11 (held auto-injector pressed fully down through second "click" sound) were checked as "yes."
Time Frame: Week 4
Population: Usability Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- M923 40 mg: Participants self-administered 40 mg of M923 every 2 weeks, as a subcutaneous injection using an auto-injector, for up to a maximum of 32 weeks.
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants
  Successfully completed P7, P10, and P11 | 31
  Successfully completed all 14 instructions | 31

3. Secondary Outcome: Number of Participants With Hazard-free Injections as Assessed by the Observer at Week 4
Description: Observers assessed usability by using a potential hazard checklist. If all potential hazards in the checklist were checked as "no," the assessment was coded as hazard free.
Time Frame: Week 4
Population: Usability Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants | 31

4. Secondary Outcome: Usability of the Auto-injector at Baseline
Description: The usability measure was the participant rating captured in the PRE- and POST- SIAQ modules at Baseline. The PRE-SIAQ module is a 7-item questionnaire that investigates feelings about injections, self-confidence (regarding self-administration), and satisfaction with self-injection. The POST-SIAQ module is a 27-item questionnaire that assesses feelings about injections, self-image, self-confidence (regarding self-administration), pain and skin reactions during or after injection (injection-site reactions), ease of use of the self-injection device, and satisfaction with self-injection. Participants rated each item of the SIAQ on a 5-point (or 6-point) semantic Likert-type scale, where a score of 1 corresponds to a participant's worst experience and a score of 5 (or 6) corresponds to a participant's best experience. Item scores were transformed to obtain a score ranging from 0 (worst experience) to 10 (best experience) for each item.
Time Frame: Baseline (Day 1)
Population: Usability Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Scores on a scale
  Feelings about injections: PRE | 7.20 (2.810)
  Feelings about injections: Post | 7.98 (2.507)
  Self-image: POST | 9.52 (1.357)
  Self-confidence: PRE | 6.34 (3.218)
  Self-confidence: POST | 7.96 (2.535)
  Pain/skin reactions: POST | 8.99 (0.865)
  Pain during/after injection: POST | 8.15 (1.591)
  Skin reaction: POST | 9.84 (0.326)
  Ease of use of the AI: POST | 8.26 (1.956)
  Satisfaction with AI: PRE | 7.98 (2.365)
  Satisfaction with AI: POST | 8.57 (1.490)

5. Secondary Outcome: Usability of the Auto-injector at Week 2
Description: The usability measure was the participant rating captured in the PRE- and POST- SIAQ modules at Week 2. The PRE-SIAQ module is a 7-item questionnaire that investigates feelings about injections, self-confidence (regarding self-administration), and satisfaction with self-injection. The POST-SIAQ module is a 27-item questionnaire that assesses feelings about injections, self-image, self-confidence (regarding self-administration), pain and skin reactions during or after injection (injection-site reactions), ease of use of the self-injection device, and satisfaction with self-injection. Participants rated each item of the SIAQ on a 5-point (or 6-point) semantic Likert-type scale, where a score of 1 corresponds to a participant's worst experience and a score of 5 (or 6) corresponds to a participant's best experience. Item scores were transformed to obtain a score ranging from 0 (worst experience) to 10 (best experience) for each item.
Time Frame: Week 2
Population: Usability Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Scores on a scale
  Feelings about injections: PRE | 7.82 (2.294)
  Feelings about injections: POST | 8.06 (2.057)
  Self-image: POST | 9.60 (1.307)
  Self-confidence: PRE | 7.77 (2.311)
  Self-confidence: POST | 8.09 (2.319)
  Pain/skin reactions: POST | 9.22 (0.747)
  Pain during/after injection: POST | 8.55 (1.490)
  Skin reactions: POST | 9.89 (0.213)
  Ease of use of the AI: POST | 8.49 (2.098)
  Satisfaction with AI: PRE | 8.39 (1.773)
  Satisfaction with AI: POST | 8.65 (1.448)

6. Secondary Outcome: Number of Participants With Successful Injections as Assessed by the Observer at Baseline
Description: as for outcome 2
Time Frame: Baseline (Day 1)
Population: Usability Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants
  Successfully completed P7, P10, and P11 | 31
  Successfully completed all 14 instructions | 31

7. Secondary Outcome: Number of Participants With Hazard-free Injections as Assessed by the Observer at Baseline
Description: as for outcome 3
Time Frame: Baseline (Day 1)
Population: Usability Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants | 31

8. Secondary Outcome: Number of Participants With Successful Injections as Assessed by the Observer at Week 2
Description: as for outcome 2
Time Frame: Week 2
Population: Usability Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants
  Successfully completed P7, P10, and P11 | 31
  Successfully completed all 14 instructions | 31

9. Secondary Outcome: Number of Participants With Hazard-free Injections as Assessed by the Observer at Week 2
Description: as for outcome 3
Time Frame: Week 2
Population: Usability Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants | 31

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments
Description: Hematology, clinical chemistry, and urinalysis clinical laboratory parameters were assessed. The hematology panel consisted of complete blood count, hemoglobin, hematocrit, mean cell volume, total leukocytes, and platelet counts. The clinical chemistry panel consisted of aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase, total bilirubin, lactate dehydrogenase, creatine kinase, C-reactive protein, cholesterol, triglycerides, total protein, sodium, potassium, chloride, blood urea nitrogen, creatinine, albumin, calcium, phosphate, glucose, glycosylated hemoglobin, uric acid, and bicarbonate. The urinalysis panel consisted of leucocytes, protein, bilirubin, urobilinogen, glucose, ketones, blood pH, nitrite, and specific gravity. Clinical significance was assessed by the Investigator.
Time Frame: Baseline; 32 Weeks
Population: Safety Analysis Set: all participants who received study medication
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants | 0

11. Secondary Outcome: Number of Participants With Vital Signs Outside the Expected Range
Description: Vital signs included respiratory rate, body temperature, pulse rate, and systolic and diastolic blood pressure.
Time Frame: 32 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants | 13

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Twelve-lead Electrocardiogram (ECG) Findings
Description: Clinical significance was assessed by the Investigator.
Time Frame: Baseline; 32 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants | 0

13. Secondary Outcome: Number of Participants With Adverse Events Leading to Premature Study Withdrawal
Description: The number of participants who had an adverse event that led to premature study withdrawal was assessed.
Time Frame: 32 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants | 2

14. Secondary Outcome: Number of Participants With Treatment-emergent Injection Site Reactions
Description: An injection site reaction is defined as pain, tenderness, erythema/redness, induration/swelling, and other. If an injection site reaction was observed, a physician was to characterize and document the reaction as an adverse event (AE). Treatment-emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the first dose of study medication, until study completion/withdrawal or within 30 days following the last treatment for early withdrawn participants.
Time Frame: 32 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants | 1

15. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With Evidence of Seroconversion as Measured by Titer of Anti-drug Antibodies (ADAs) at Baseline
Description: A participant was considered to have developed ADAs if a confirmed positive result was observed at any time during the treatment period post-dose (irrespective of titer value). Samples were collected predose (prior to administering investigational product) and before any hematology/chemistry samples were drawn at that visit.
Time Frame: Baseline (Day 1)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants
  Overall ADA/negative predose | 6
  Overall ADA/positive predose | 27

16. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With Evidence of Seroconversion as Measured by Titer of ADAs at Week 4
Description: as for outcome 15
Time Frame: Week 4
Population: Safety Analysis Set. Only those participants contributing data at Week 4 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 32
Participants
  Overall ADA/negative | 6
  Overall ADA/positive | 26

17. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With Evidence of Seroconversion as Measured by Titer of ADAs at Week 12
Description: as for outcome 15
Time Frame: Week 12
Population: Safety Analysis Set. Only those participants contributing data at Week 12 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 23
Participants
  Overall ADA/negative | 5
  Overall ADA/positive | 18

18. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With Evidence of Seroconversion as Measured by Titer of ADAs at Week 24
Description: as for outcome 15
Time Frame: Week 24
Population: Safety Analysis Set. Only those participants contributing data at Week 24 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 22
Participants
  Overall ADA/negative | 5
  Overall ADA/positive | 17

19. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With Evidence of Seroconversion as Measured by Titer of ADAs at the Safety Follow-Up Visit
Description: as for outcome 15
Time Frame: Safety Follow-Up Visit (32 Weeks)
Population: Safety Analysis Set. Only those participants contributing data at Week 32 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants
  Overall ADA/negative | 6
  Overall ADA/positive | 25

20. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With Neutralizing Anti-drug Antibodies (nADAs) at Baseline
Description: A participant was considered to have developed nADAs if a confirmed positive result was observed at any time during the treatment period post-dose. Samples were collected predose (prior to administering investigational product) and before any hematology/chemistry samples were drawn at that visit.
Time Frame: Baseline (Day 1)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 33
Participants
  Overall nADA/negative | 26
  Overall nADA/positive | 7

21. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With nADAs at Week 4
Description: as for outcome 20
Time Frame: Week 4
Population: Safety Analysis Set. Only those participants contributing data at Week 4 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 32
Participants
  Overall nADA/negative | 26
  Overall nADA/positive | 6

22. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With nADAs at Week 12
Description: as for outcome 20
Time Frame: Week 12
Population: Safety Analysis Set. Only those participants contributing data at Week 12 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 23
Participants
  Overall nADA/negative | 17
  Overall nADA/positive | 6

23. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With nADAs at Week 24
Description: as for outcome 20
Time Frame: Week 24
Population: Safety Analysis Set. Only those participants contributing data at Week 24 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 22
Participants
  Overall nADA/negative | 18
  Overall nADA/positive | 4

24. Secondary Outcome: Immunogenicity of M923 Assessed as the Number of Participants With nADAs at the Safety Follow-Up Visit
Description: as for outcome 20
Time Frame: Safety Follow-Up Visit (32 Weeks)
Population: Safety Analysis Set. Only those participants contributing data at Week 32 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M923 40 mg
Number analyzed (Participants) | 31
Participants
  Overall nADA/negative | 24
  Overall nADA/positive | 7

ADVERSE EVENTS:
Time Frame: From the date of Screening until the Safety Follow-Up Visit (approximately 32 weeks)
Description: Safety Analysis Set: all participants who received study medication
Arm/Group | M923 40 mg
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M923 40 mg (N=33)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M923 40 mg (N=33)
Administrative site pain (General disorders) | 2
Injection site bruising (General disorders) | 5
Injection site coldness (General disorders) | 4
Injection site erythema (General disorders) | 10
Injection site induration (General disorders) | 2
Injection site pain (General disorders) | 27
Injection site pruritus (General disorders) | 4
Injection site swelling (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT02722044/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT02722044/SAP_001.pdf